CLINICAL TRIAL: NCT01694147
Title: Extravascular Lung Water Index Exhibits Pulmonary and Systemic Permeability in Patients With Sepsis Related Acute Lung Injury/Acute Respiratory Distress Syndrome.
Brief Title: EVLWI Exhibits Pulmonary and Systemic Permeability in Sepsis Related ALI/ARDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chung Fu-Tsai, Attending physician, Chang Gung Memorial Hospital
Other Study IDs: 99-3957B
Record Dates: First submitted 2012-09-23; First posted 2012-09-27 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2012-09

CONDITIONS: Sepsis Related Acute Lung Injury/Acute Respiratory Distress Syndrome
Keywords: relationship; endothelial injury; vascular permeability; severe sepsis related ALI/ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — To measure the relationship between endothelial injury (serum TM, vWF, VEGF, TIE-2 increase and imbalance of ANG-1/ANG-2) and vascular permeability and EVLWI in patients, 20ml peripheral blood will be sampling retented on day 1 and day 3 after including.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients with sepsis related ALI/ARDS.: Consecutive septic patients with ALI/ARDS in medical intensive care units (ICUs) will be enrolled. EVLWI will be measured by PiCCO monitoring system.
  Interventions: Device: PiCCO monitoring system

INTERVENTIONS:
Device: PiCCO monitoring system — The EVLW measurement will be based on transpulmonary thermodilution method. This method was recently introduced as part of the PiCCO plus system (Pulsion Medical System, Munich, Germany), for monitoring severe sepsis patients being treated in medical ICUs. This method only used a single indicator (cold saline solution), and demonstrated a satisfactory correlation with the gravimetric method. A 4-F arterial catheter (PulsiocathPV2014L16; Pulsion Medical Systems, Munich, Germany) was positioned in the descending aorta via the femoral artery using the Seldinger technique. The femoral arterial catheter and a standard central venous catheter were connected to pressure transducers, and also to an integrated bedside monitor (PiCCO; Pulsion Medical Systems).

SUMMARY:
To investigate the possible mechanisms of pulmonary and systemic permeability change including cytokine, extravascular lung water index (EVLWI), and oxygenation parameters in patients with sepsis related acute lung injury (ALI)/acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
This investigation is a prospective control study. Informed consents will be obtained from all patients or their surrogates prior to the procedure of EVLWI measurement and blood sampling for molecular measurement including cytokines.

From July 2011 to June 2014, consecutive septic patients with ARDS in intensive care units (ICUs) will be enrolled at Chang Gung Memorial Hospital, a university-affiliated hospital in Taiwan. EVLWI will be measured by PiCCO monitoring system. Serum cytokine such as endothelin-1, TNF-alfa, IL-6, Tie-1, Tie-2, angiopoietin-1, angiopoietin-2,VEGF and thrombomodulin will be measured.

ELIGIBILITY:
Inclusion Criteria:

* sepsis in ICU within 48 hours,
* mechanical ventilator use,
* PaO2/FiO2 < 300,

Exclusion Criteria:

* age younger than 20 years,
* known pregnancy,
* participation in another trial within 30 days before meeting the eligibility criteria, and
* terminal malignancy.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Septic patients receiving endotracheal mechanical ventilation for hypoxemic acute respiratory failure were eligible if the following criteria were met for no more than 48 hours before enrollment: ratio of partial pressure of arterial oxygen over fraction of inspired oxygen (PaO2:FIO2) no greater than 300 mm Hg at time of enrollment, recent appearance of bilateral pulmonary infiltrates consistent with edema, and no clinical evidence of left atrial hypertension (pulmonary-capillary wedge pressure _18 mm Hg, when available).
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-07; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
vascular permeability of sepsis related ALI/ARDS | 3 days
  vascular permeability (day 1 and 3 EVLWI, lung permeability, 24hr fluid balance, microalbuminuria, DAMPs/RAGE, Ang-1, 2 and TIE-2 level, will be detected in the blood sampling) and sepsis-induced ALI/ARDS.

SECONDARY OUTCOMES:
relationship between endothelial injury and vascular permeability. | 3 days
  relationship between endothelial injury (serum TM, vWF, VEGF, TIE-2 increase and imbalance of ANG-1/ANG-2) and vascular permeability in patients with sepsis related ALI/ARDS.

CONTACTS AND LOCATIONS:
Locations (1):
- Chung Gung Memorial Hospital, Linkou, Taiwan, Taiwan